CLINICAL TRIAL: NCT03348020
Title: Iron Homeostasis, Adipose Tissue Lipolysis, and Insulin Resistance in Overweight and Obese Humans
Brief Title: Iron and Insulin Resistance in Overweight and Obese Humans
Acronym: Fe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science and Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00138926
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Glucose Intolerance; Insulin Resistance; Iron Metabolism
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Clinical Trial (Experimental): Before blood donation, subjects will participate in a baseline clinical trial where the research team will perform a series of metabolic tests as described in the detailed study description.
  Interventions: Procedure: Blood Donation
- Post-Blood Donation Clinical Trial (Experimental): 1 month after blood donation, subjects will participate in post-blood donation clinical trial where the research team will perform a series of metabolic tests as described in the detailed study description.
  Interventions: Procedure: Blood Donation

INTERVENTIONS:
Procedure: Blood Donation — Subjects will donate blood within ~1 month after their baseline clinical trial. Subjects will report to the Substrate Metabolism Laboratory between 24 and 72 hours following blood donation. A finger-stick will be performed for the measurement of hemoglobin concentration.

SUMMARY:
Determine the effects of reducing whole-body iron stores in overweight/obese subjects (via one-time blood donation) on adipose tissue iron content, factors regulating iron homeostasis and lipolytic rate in adipose tissue, as well as measures of adipose tissue and whole-body insulin resistance.

After a screening visit to determine eligibility, subjects will undergo a battery of tests for the determination of primary outcome measures at baseline. They will then donate 1 unit (~500 mL) of blood (at a local blood donation center) and return for a follow-up testing 4 weeks after blood donation. During the 4-week period between study trials, subjects will be required to maintain a stable body mass and not alter their dietary or physical activity habits.

DETAILED DESCRIPTION:
Screening:

If a potential subject meets the eligibility criteria after completing the general pre-screening questionnaire, they will be contacted to set up an in-person screening visit where the comprehensive written informed consent will be obtained. This visit may occur either at the Michigan Clinical Research Unit (MCRU) or at the Substrate Metabolism Laboratory (SML). Subjects will complete health history, food frequency, and physical activity questionnaires. Subjects that meet eligibility requirements and provide written informed consent will have a finger-stick performed for the assessment of hemoglobin concentration. Women with hemoglobin < 13.0 g/dL and men with hemoglobin < 14.0 g/dL will be withdrawn from the study.

Percent body fat will be measured using Dual Energy X-ray Absorptiometry [DEXA]. Women will provide a urine sample for a urine pregnancy test prior to the DEXA scan; if a subject has a positive pregnancy test prior to the DEXA scan, they will be withdrawn. The DEXA body composition assessment test may be performed at the screening visit or scheduled anytime between the screening visit and the baseline trial.

Baseline Trial:

Subjects will be provided general instructions on what to eat in the 3 days leading up to their baseline trial and be required to abstain from planned exercise in the 3 days leading up to the baseline and post-blood donation study trials. They will record their dietary intake during the 3 days leading up to the baseline trial and replicate it during the 3 days prior to the post-blood donation study trial. They will be required to fast the night before the trials starting at 9:00PM.

Subjects will arrive at MCRU at ~07:00AM. After measurement of body weight and resting blood pressure, intravenous catheters (IV) will be placed in each arm (one for blood sampling and the other for infusion).

At ~7:50 AM blood samples (in 5 minute intervals) will be collected. A ~8:00 AM a tracer-labeled glycerol infusion will begin. The tracer-labeled glycerol infusion that is infused occurs naturally in the body. By injecting a slightly greater amount of this substance than is already in the body, the rate of fat breakdown and fat burning is able to be measured. One of the subject's hands will be placed within a "hot-hand box" to enable the study team to collect arterialized venous blood samples from the intravenous catheter. At ~08:30AM, a small sample of abdominal fat tissue will be collected. Between ~09:50 and 10:00, three blood samples will be collected to determine basal lipolysis. At ~10:00, we will start the hyperinsulinemic, euglycemic clamp procedure to measure the body's sensitivity to insulin. During this procedure insulin and glucose will be infused through the IV in the forearm and blood samples will be collected periodically to monitor the subjects blood sugar. The infusion rate of glucose will be changed accordingly to ensure that the subjects blood sugar is maintained at a healthy/normal level. This procedure will take about two hours. Following completion, The insulin will be discontinued and the subject will be provided a lunch and the glucose will be gradually tapered off over the next hour. The study team will ensure the subjects blood glucose levels are stable prior to discharge.

Blood Donation:

Subjects will donate blood within ~1 month after their baseline trial. Subjects will report to the Substrate Metabolism Laboratory between 24 and 72 hours following blood donation. A finger-stick will be performed for the measurement of hemoglobin concentration.

Post-Blood Donation Trial:

The exact same procedures as performed in the Baseline Trial will be repeated 4 weeks after the subject's blood donation.

Diet/Physical Activity/Weight Maintenance:

Subjects will be required to maintain their normal diet and physical activity habits during the study. Following the baseline trial, subjects will be provided with a scale and asked to weigh themselves at home on a daily basis. If body weight changes ±2kg from their initial weight, subjects will consult with our research dietitian for strategies to maintain weight during the period between study trials.

ELIGIBILITY:
Subject Inclusion Criteria

* Age: 18-40
* (Body Mass Index ≥27 kg/m2>27)
* Women must have regularly occurring menses and must be premenopausal
* Meet general blood donation eligibility requirements

Subject Exclusion Criteria

* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism, or inflammation
* Blood donation in the last 12 months
* Iron supplementation in the last 12 months (multivitamin with ≤100 %DV ok)
* Diagnosed anemia in the last 24 months
* Weight instability ≥ ±3kg in the last 6 months
* Women must not be pregnant or actively lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity after blood donation | 1 month
  A hyperinsulinemic-euglycemic clamp will be used to assess insulin sensitivity. The change in the glucose infusion rate will be used to measure the insulin sensitivity after blood donation.

SECONDARY OUTCOMES:
Change in lipolytic rate after blood donation | 1 month
  rate of appearance of glycerol

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Horowitz, Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No